CLINICAL TRIAL: NCT06296212
Title: Multicenter, Randomized, Double-blind, Phase III Study of Intravenous TAD® 600 Mg/4 ML Solution for Injection to Evaluate Efficacy and Safety in Preventing Myocardial Injury in Patients with Pneumonia.
Brief Title: Study of Intravenous TAD® 600 Mg/4 ML Solution for Injection to Evaluate Efficacy and Safety in Preventing Myocardial Injury in Patients with Pneumonia.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biomedica Foscama S.p.A. Industria Chimico-Farmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GLT-07-22
Record Dates: First submitted 2024-02-27; First posted 2024-03-06 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-07

CONDITIONS: Pneumonia; Myocardial Injury
MeSH Terms: conditions — Pneumonia | interventions — DAT protocol 1; Powders; Solvents; Solutions; Injections; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAD® 600 mg/4 mL Solution for Injection (Experimental): TAD® 600 mg/4 mL powder and solvent for solution for injection, 1 vial powder (glutathione sodium salt 646 mg) + 1 solvent ampoule (4 mL water for injection) reconstituted solution in 50 mL of 0.9% sodium chloride solution) administered intravenously (with an infusion rate of 10 mL/min), 2 times a day (with a dosing interval of 8 hours ± 30 minutes) for 5 consecutive days (Day 1, Day 2, Day 3, Day 4 and Day 5). Doses will be administered at the same time of the day (every 24 hours ± 30 minutes).
  Interventions: Drug: TAD® 600 mg/4 mL powder and solvent for solution for injection
- Saline solution of 0.9% sodium chloride (Placebo Comparator): Placebo (50 mL of 0.9% sodium chloride solution) administered intravenously (with an infusion rate of 10 mL/min), 2 times a day (with a dosing interval of 8 hours ± 30 minutes) for 5 consecutive days (Day 1, Day 2, Day 3, Day 4 and Day 5). Doses will be administered at the same time of the day (every 24 hours ± 30 minutes).
  Interventions: Drug: Saline solution 0.9% of sodium chloride

INTERVENTIONS:
Drug: TAD® 600 mg/4 mL powder and solvent for solution for injection — TAD® 600 mg/4 mL powder and solvent for solution for injection, 1 vial powder (glutathione sodium salt 646 mg) + 1 solvent ampoule (4 mL water for injection) reconstituted solution in 50 mL of 0.9% sodium chloride solution) administered intravenously (with an infusion rate of 10 mL/min), 2 times a day (with a dosing interval of 8 hours ± 30 minutes) for 5 consecutive days (Day 1, Day 2, Day 3, Day 4 and Day 5). Doses will be administered at the same time of the day (every 24 hours ± 30 minutes).
  Arms: TAD® 600 mg/4 mL Solution for Injection
Drug: Saline solution 0.9% of sodium chloride — Placebo (50 mL of 0.9% sodium chloride solution) administered intravenously (with an infusion rate of 10 mL/min), 2 times a day (with a dosing interval of 8 hours ± 30 minutes) for 5 consecutive days (Day 1, Day 2, Day 3, Day 4 and Day 5). Doses will be administered at the same time of the day (every 24 hours ± 30 minutes).
  Arms: Saline solution of 0.9% sodium chloride

SUMMARY:
The goal of this PHASE III clinical trial is to evaluate efficacy and safety of intravenous TAD® 600 mg/4 mL solution for injection in preventing myocardial injury in patients with pneumonia.

The main question it aims to answer is:

• could TAD® used as an add-on treatment to the standard therapy, due to the presence of the sodium salt glutathione, be effective and safe in preventing the risk of developing myocardial injury in hospitalized patients with pneumonia?

Patients diagnosed with pneumonia (in the emergency department or hospital ward) will be asked to participate in the study and sign the Informed Consent Form (ICF) to assess their eligibility for enrollment.

Eligible patients who meet the study inclusion criteria and complete the required Screening & Baseline (V0) examinations, will be randomized with a 1:1 ratio allocation to the IMP Test group (TAD® treatment) or IMP Placebo group (Placebo treatment) in a double-blind manner, PI & Patient blinded.

TAD® (600 mg/4 mL reconstituted solution in 50 mL of 0.9% sodium chloride solution) or Placebo (50 mL of 0.9% sodium chloride solution) will be administered:

* intravenously (with an infusion rate of 10 mL/min)
* 2 times a day (with a dosing interval of 8 hours ± 30 minutes)
* for 5 consecutive days (Day 1, Day 2, Day 3, Day 4 and Day 5)
* patients will then be required to undergo five Follow-up Visits.

ELIGIBILITY:
Inclusion Criteria

* Patients with an age of ≥ 18 and ≤ 80 years
* Diagnosis of CAP or HAP requiring hospitalization
* Patients with one of the following :

  - At least one cardiovascular comorbidity:
* Chronic atrial fibrillation
* History of ischemic heart disease (≥ 3 months)
* Heart failure
* Cardiac Valvular Disease
* Previous (≥ 6 months) episode of myocarditis or pericarditis.

  - Very high risk of developing cardiovascular diseases according to the SCORE2 and SCORE2-OP risk models for moderate risk European regions (score ≥ 7.5% for patients < 50 years old, score ≥ 10% for patients 50-69 years old, and score ≥ 15% for patients ≥ 70 years old).
* Provision of written informed consent as approved by the Ethics Committee (EC).

Exclusion Criteria

Medical Conditions:

* Active malignancy
* Severe heart failure (NYHA class III and IV)
* End-stage renal failure (eGFR < 30 mL/min)
* Severe liver disease
* History of hypersensitivity to glutathione or any excipients
* Use of drugs containing sacubitril
* Use of drugs with antioxidant activity in the last 3 months
* Use of narcotics
* Use of invasive mechanical ventilation
* Recent (< 3 months) ACS (STEMI, NSTEMI, UA), myocardial revascularization, myocarditis, acute pericarditis episodes.

General Conditions:

* Pregnant or breastfeeding women
* Women of child-bearing potential not using at least one effective contraceptive method for the entire trial
* Participation in other investigational drug or device clinical trials within 30 days prior to study screening
* Patients legally or mentally incapacitated unable to give informed consent for the participation in this trial
* Patients unable or unwilling to comply with the appointments after hospitalization or with all the requirements of the Protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of the change of levels of high-sensitivity cardiac Troponin (hs-cTn) at V1 versus V0 in the two groups. | 7-9 days
  Change of levels of high-sensitivity cardiac Troponin (hs-cTn) between V1 and V0 will be calculated. The non-paired T test or Mann Whitney test will be used to compare changes between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Noemi Evangelisti, Study Director — Biomedica Foscama S.p.A
Locations (7):
- Italy (7):
  - Azienda Ospedaliero-Universitaria Pisana, Pisa, PI
  - Fondazione Policlinico Universitario Campus Bio-Medico, Roma, RM
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Roma, RM
  - Azienda Ospedaliero-Universitaria Policlinico Umberto I, Roma, RM
  - Azienda Ospedaliero-Universitaria Sant'Andrea, Roma, RM
  - Azienda Ospedaliera Santa Maria, Terni, TR
  - Ospedale Ca' Foncello, Treviso, TV

IPD SHARING:
Plan to Share IPD: No